CLINICAL TRIAL: NCT02684760
Title: A Phase 1, Open Label, Single-dose 3-way Crossover Study To Evaluate The Relative Bioavailability Of A Solid Dose Formulation Of Pf-06651600 Under Fasting Conditions And The Effect Of A High Fat Meal On The Bioavailability Of The Solid Dosage Formulation Of Pf-06651600 In Healthy Subjects
Brief Title: Bioavailability Study Of PF-06651600 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981003; 2015-004857-41 (EudraCT Number)
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — PF-06651600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1: PF-06651600 (Experimental): Single dose of PF-06651600 50 mg tablet (under fasted condition and following high fat meal) and 50 mg oral formulation (under fasted condition) to evaluate bioavailability.
  Interventions: Drug: PF-06651600
- Cohort 2: PF-06651600 (Experimental): Single dose of PF-06651600 50 mg tablet (under fasted condition and following high fat meal) and 50 mg oral formulation (under fasted condition) to evaluate bioavailability.
  Interventions: Drug: PF-06651600
- Cohort 3: PF-06651600 (Experimental): Single dose of PF-06651600 50 mg tablet (under fasted condition and following high fat meal) and 50 mg oral formulation (under fasted condition) to evaluate bioavailability.
  Interventions: Drug: PF-06651600
- Cohort 4: PF-06651600 (Experimental): Single dose of PF-06651600 50 mg tablet (under fasted condition and following high fat meal) and 50 mg oral formulation (under fasted condition) to evaluate bioavailability.
  Interventions: Drug: PF-06651600
- Cohort 5: PF-06651600 (Experimental): Single dose of PF-06651600 50 mg tablet (under fasted condition and following high fat meal) and 50 mg oral formulation (under fasted condition) to evaluate bioavailability.
  Interventions: Drug: PF-06651600
- Cohort 6: PF-06651600 (Experimental): Single dose of PF-06651600 50 mg tablet (under fasted condition and following high fat meal) and 50 mg oral formulation (under fasted condition) to evaluate bioavailability.
  Interventions: Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 — PF-06651600 will be administered as a tablet and extemporaneously prepared solution in each cohort.

SUMMARY:
PF-06651600 is being developed for treatment of inflammatory bowel disease. This study will test the bioavailability of a solid dose formulation of PF-06651600 compared to an oral solution formulation under fasting conditions and the effect of a high fat meal on the bioavailability of the solid dose formulation of PF-06651600 in healthy subjects. Safety and tolerability of the tablet and oral solution formulations of PF-06651600 will be assessed under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female subjects between 18 and 55 years old, inclusive. Females must be of non-child bearing potential.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Prior history of chicken pox.
* Evidence of personally signed and dated informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, lab tests and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, GI, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males.
* Screening blood pressure >140/90 mm Hg.
* Screening laboratory abnormalities as defined by the protocol.
* Unwilling or unable to comply with the Lifestyle Guidelines as defined by the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-06651600 | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06651600 | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Cmax) for PF-06651600 | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Plasma Decay Half Life (t1/2) for PF-06651600 | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Time to Reach Maximum Concentration (Tmax) for PF-06651600 | 0, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Time to Reach Maximum Concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Saadeddin A, Purohit V, Huh Y, Wong M, Maulny A, Dowty ME, Sagawa K. Virtual Bioequivalence Assessment of Ritlecitinib Capsules with Incorporation of Observed Clinical Variability Using a Physiologically Based Pharmacokinetic Model. AAPS J. 2024 Jan 24;26(1):17. doi: 10.1208/s12248-024-00888-9. PMID 38267790
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Purohit V, Huh Y, Wojciechowski J, Plotka A, Salts S, Antinew J, Dimitrova A, Nicholas T. Leveraging Prior Healthy Participant Pharmacokinetic Data to Evaluate the Impact of Renal and Hepatic Impairment on Ritlecitinib Pharmacokinetics. AAPS J. 2023 Mar 28;25(3):32. doi: 10.1208/s12248-023-00792-8. PMID 36977960
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981003&StudyName=A+Phase+1%2C+Open+Label%2C+Single-dose+3-way+Crossover+Study+To+Evaluate+The+Relative+Bioavailability+Of+A+Solid+Dose+Formulation+Of+Pf-06651600+Under+Fasting+Conditions+And+The+Effect+Of+A+High+Fat+Meal+On+The+Bioavailability+Of+The+Solid+Dosage+Formulation+Of+Pf-06651600+In+Healthy+Subjects